CLINICAL TRIAL: NCT02932748
Title: Weight Management in Rural Communities
Acronym: M-DEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSCL03396; R01DK108732 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-10-13 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Weight Loss; Obesity; Body Weight
MeSH Terms: conditions — Weight Loss; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group Phone Conference Call (Experimental): Delivery: Group Phone Diet: PCMs
  Interventions: Dietary Supplement: Portion Controlled Meals (PCM); Behavioral: Group Phone (GP)
- Individual Phone Call (Experimental): Delivery: Individual Phone Call Diet: PCMs
  Interventions: Dietary Supplement: Portion Controlled Meals (PCM); Behavioral: Individual Phone (IP)
- Enhanced Usual Care (Active Comparator): Delivery: Face-to-Face Diet: Conventional Diet
  Interventions: Dietary Supplement: Conventional Diet; Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Dietary Supplement: Portion Controlled Meals (PCM) — Portion controlled meals provide conveniently packaged, low-energy, high-nutritional content food.
  Arms: Group Phone Conference Call; Individual Phone Call
Behavioral: Group Phone (GP) — Weight management program delivered via group conference call.
  Arms: Group Phone Conference Call
Dietary Supplement: Conventional Diet — Conventional diet (CD) will consist of a nutritionally balanced, reduced energy, high volume, lower fat (fat= 20-30% energy) diet based on USDA's MyPlate recommendations.
  Arms: Enhanced Usual Care
Behavioral: Individual Phone (IP) — Weight management program delivered via individual phone call.
  Arms: Individual Phone Call
Behavioral: Enhanced Usual Care (EUC) — Weight management topics delivered face-to-face at clinic office every 6 months.
  Arms: Enhanced Usual Care

SUMMARY:
The goal of this study is to evaluate the effect of three weight management interventions (group phone conference calls, individual phone calls, and enhanced usual care) on weight across 18 months in overweight and obese adults recruited through and treated by rural primary care clinics.

DETAILED DESCRIPTION:
The rates of overweight/obesity are significantly higher among residents of rural areas compared to their urban counterparts. Recent focus to provide whole-person health care suggests that rural primary care clinics may provide an ideal setting for delivery of weight management.

This study is a 3 group randomized trial to evaluate intervention delivery. The investigators will randomize 200 overweight/obese adult residents of rural towns (town population < 50,000) who obtain health care at primary care clinics to one of three groups for an 18 month trial (6 month weight loss; 12 month weight maintenance).

Group 1) Group phone (GP)/Portion-Controlled Meals (PCM)

Group 2) Individual phone (IP)/PCM

Group 3) Enhanced usual care (EUC)/Conventional Diet (CD)

All participants will receive a progressive physical activity program. Physical activity will progress from 45 min/wk in month 1 to 225 min/wk in month 4 and remain at 225 min/wk for the duration of the 18 month study for Group 1 & 2. Physical activity will progress from 45 min/wk in month 1 to 150 min/wk in month 4 and remain at 150 min/wk for the duration of the 18 month study for Group 3.

Participants on the CD will be asked to consume a nutritionally balanced, reduced energy, high volume, lower fat (fat= 20-30% energy) diet recommended by the Academy of Nutrition and Dietetics and the USDA's MyPlate approach. Examples of meal plans consisting of suggested servings of proteins, grains, fruits and vegetables, dairy and fats based on individuals energy needs will be provided. Participants using PCM will consume PCMs with the addition of 5 fruits and vegetables per day during weight loss.

EUC will meet with a health educator every 6 months to discuss weight management topics. GP & IP will receive the weight management intervention over the phone weekly during weight loss and biweekly during weight maintenance tracking diet and physical activity and will submit the results to a health educator prior to every meeting.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25 to 45 kg/m2
* Clearance from primary care physician

Exclusion Criteria:

* Unable to participate in moderate intensity physical activity
* Participation in weight loss or physical activity program in previous 6 months
* Greater than 3, 30-min bouts of planned exercise/week
* Not weight stable (+/-4.6 kg) for 3 months prior to intake
* Unwilling to be randomized to 1 of the 3 study groups
* Report being pregnant during the previous 6 months or planned pregnancy in the following 18 months
* Serious medical risk such as cancer, recent cardiac event
* Current use of antipsychotics or untreated depression
* Adherence to specialized diet regimens (food allergy, vegetarian, macrobiotic)
* Binge eating disorder
* Planning to movie to a location and no longer having access to rural clinic site

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, EdD, Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Derived] Gorczyca AM, Washburn RA, Ptomey LT, Mayo MS, Krebill R, Sullivan DK, Gibson CA, Stolte S, Donnelly JE. Weight management in rural health clinics: Results from the randomized midwest diet and exercise trial. Obes Sci Pract. 2024 Apr 24;10(2):e753. doi: 10.1002/osp4.753. eCollection 2024 Apr. PMID 38660371
- [Derived] Gorczyca AM, Washburn RA, Ptomey L, Mayo MS, Sullivan DK, Gibson CA, Lee R, Stolte S, Donnelly JE. Weight management in rural health clinics: The Midwest diet and exercise trial. Contemp Clin Trials. 2018 Apr;67:37-46. doi: 10.1016/j.cct.2018.02.006. Epub 2018 Feb 15. PMID 29454140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Started | 71 | 80 | 36
Completed | 47 | 60 | 28
Not Completed | 24 | 20 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care | Total
Number analyzed (Participants) | 71 | 80 | 36 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.2) | 49.4 (11.2) | 50.4 (13.8) | 50.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 66 | 28 | 153
  Male | 12 | 14 | 8 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 62 | 70 | 32 | 164
  Unknown or Not Reported | 8 | 9 | 4 | 21
Region of Enrollment [Number; unit: participants]
  United States | 71 | 80 | 36 | 187
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.6 (4.7) | 34.6 (4.5) | 35.2 (4.5) | 35.1 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Change Over 6 Months
Description: Mean weight change (kg) of participants between the three study groups.
Time Frame: Change in baseline to 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 47 | 60 | 28
kilograms | -11.4 (6.7) | -9.1 (6.8) | -2.6 (4.8)
Statistical Analysis 1: Comparison: Group Phone Conference Call vs Individual Phone Call vs Enhanced Usual Care; Test type: Superiority; p < .0001, ANOVA — A global one-way ANOVA was followed by two pairwise t-tests on the comparisons of interest, i.e., IP vs. EUC, and GP vs IP for weight change across 6 months, evaluated at p ≤ 0.025, using both intent-to-treat and completer only data

2. Secondary Outcome: Change in BMI Across 6 Months
Description: Mean BMI change (kg/m^2) of participants between the three study groups.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 47 | 60 | 28
kg/m^2 | -4.1 (2.2) | -3.2 (2.3) | -0.9 (1.6)

3. Secondary Outcome: Change in Waist Circumference Across 6 Months
Description: Mean waist circumference change (cm) in the three study groups.
Time Frame: Change from baseline - 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 45 | 60 | 28
cm | -7.2 (6.1) | -6.1 (5.8) | -2.1 (4.5)

4. Secondary Outcome: Triglycerides
Description: Mean change in fasting triglycerides will be compared across all treatment arms.
Time Frame: Change from baseline to 6 months
Population: Blood values were missing for n=2 in GP, n=7 in IP and n=2 in EUC.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 43 | 53 | 26
mg/dL | -26.2 (39) | -29.4 (61.3) | 4.8 (39.1)

5. Secondary Outcome: HDL-cholesterol
Description: Mean change in fasting HDL-cholesterol will be compared across all treatment arms.
Time Frame: Change from baseline to 6 months
Population: Blood values were missing for n=2 in GP, n=7 in IP and n=2 in EUC.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 43 | 53 | 26
mg/dL | 0.3 (9.6) | 0.3 (9.6) | 1.6 (6.2)

6. Secondary Outcome: Change in Systolic Blood Pressure Across 6 Months
Description: Mean change in systolic blood pressure will be compared across all treatment arms.
Time Frame: Change from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 45 | 60 | 28
mmHg | -8.6 (13.1) | -7.9 (13.4) | 1.7 (19.5)

7. Secondary Outcome: Change in Fasting Glucose Across 6 Months
Description: Mean change in fasting glucose will be compared across all treatment arms.
Time Frame: Change from baseline to 6 months
Population: Blood values were missing for n=2 in GP, n=7 in IP and n=2 in EUC.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
Number analyzed (Participants) | 43 | 51 | 26
mg/dL | -5.9 (9.7) | -4.4 (26.2) | 1.6 (8.3)

8. Secondary Outcome: Cost Effectiveness at 6 Months
Description: Cost effectiveness was calculated for the group as the average total cost of the intervention arm (GP or IP) divided by the average weight loss at 6 months of the intervention arm. Costs associated with delivering the 6-month weight loss intervention, including supplies and intervention implementation, were estimated in 2019 U.S. dollars. Supply costs, i.e., pedometers, participant notebooks, providing and shipping low-calorie shakes and printed materials for the GP and IP arms. Implementation costs, i.e., time devoted to interventionist training, preparation and delivery of behavioral sessions and email contacts with participants were estimated as the time spent in these activities obtained from interventionist time sheets multiplied by interventionists hourly wage. Due to the cost effectiveness outcome measure being a ratio between two random variables, there are no dispersion/precision measures reported.
Time Frame: 6 months
Population: Data not collected for the Enhanced Usual Care Arm/Group as this was the comparator.
Measure: Number; unit: $/kg
Arm/Group | Group Phone Conference Call | Individual Phone Call
Number analyzed (Participants) | 47 | 60
$/kg | 60 | 93

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Group Phone Conference Call | Individual Phone Call | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/80 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/80 | 1/36
Other Adverse Events (participants affected / at risk) | 0/71 | 0/80 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Phone Conference Call (N=71) | Individual Phone Call (N=80) | Enhanced Usual Care (N=36)
Cancer, breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/48/NCT02932748/Prot_SAP_000.pdf